CLINICAL TRIAL: NCT04431726
Title: A Phase IIIb, Multicenter, Open-Label, Single-Arm Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Emicizumab in Patients From Birth to 12 Months of Age With Hemophilia A Without Inhibitors
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Emicizumab in Participants From Birth to 12 Months of Age With Hemophilia A Without Inhibitors
Acronym: HAVEN 7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO41787; 2020-001733-12 (EudraCT Number); 2023-505964-13-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Severe Hemophilia A
Keywords: Severe hemophilia A Without Factor VIII Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Emicizumab (Experimental)
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Initially, all participants will receive 4 loading doses of 3 milligrams per kilogram (mg/kg) emicizumab subcutaneously (SC) once every week (QW) for 4 weeks followed by the maintenance dosing regimen 3 mg/kg emicizumab SC once every 2 weeks (Q2W) for a total of 52 weeks. Starting from Week 17 of treatment, individual participants may have their dose up-titrated to 3 mg/kg SC QW if they experience suboptimal bleeding control.
  At the Week 53 clinic visit following consultation with the treating physician, parents/caregivers may elect for their child to continue with the maintenance 3-mg/kg SC Q2W dosing regimen or to switch to the maintenance 1.5-mg/kg SC QW or 6-mg/kg SC once every 4 weeks (Q4W) dosing regimen for the subsequent 7-year long-term follow-up period.
  During the study, participants will be treated with emicizumab until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria specified in the protocol, whichever occurs first.
  Other Names: Hemlibra; RO5534262; RG6013; ACE910

SUMMARY:
This is a Phase IIIb, multicenter, open-label, single-arm study of prophylactic emicizumab in previously untreated and minimally treated patients at study enrollment from birth to ≤12 months of age with severe hemophilia A (intrinsic factor VIII [FVIII] level <1%) without FVIII inhibitors. The study is designed to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of emicizumab administered at 3 milligrams per kilogram of body weight (mg/kg) once every 2 weeks (Q2W) for 52 weeks. After 1 year of treatment, participants will continue to receive emicizumab (1.5 mg/kg once every week [QW], 3 mg/kg Q2W or 6 mg/kg once every 4 weeks [Q4W]) over a 7-year long-term follow-up period under this study frame.

ELIGIBILITY:
Inclusion Criteria:

* Age from birth to ≤12 months at time of informed consent
* Body weight ≥3 kilograms (kg) at time of informed consent. Patients with a lower body weight can be enrolled after they have reached a body weight of 3 kg. Premature babies (gestational age <38 weeks) may be enrolled as long as they have reached a body weight of 3 kg. For premature babies, the corrected gestational age should be reported.
* Mandatory receipt of vitamin K prophylaxis according to local standard practice
* Diagnosis of severe congenital hemophilia A (intrinsic FVIII level <1%)
* A negative test for FVIII inhibitor (i.e., <0.6 Bethesda units [BU]/mL) locally assessed during the 2-week screening period
* No history of documented FVIII inhibitor (i.e., <0.6 BU/mL), FVIII drug-elimination half-life <6 hours, or FVIII recovery <66%
* Previously untreated patients or minimally treated patients (i.e., up to 5 days of exposure with hemophilia-related treatments, such as plasma-derived FVIII, recombinant FVIII, fresh frozen plasma, cryoprecipitate, or whole blood products)
* Documentation of the details of the hemophilia-related treatments received since birth
* Documentation of the details of the bleeding episodes since birth
* For patients from birth to <3 months of age at the time of study entry: no evidence of active intracranial hemorrhage, as confirmed by a negative cranial ultrasound at screening irrespective of delivery mode
* Adequate hematologic, hepatic, and renal function, as defined in the protocol
* For parents/caregivers: willingness and ability to comply with the study protocol requirements, scheduled visits, treatment plans, laboratory tests, completion of applicable questionnaires, and other study procedures

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than severe hemophilia A
* Use of systemic immunomodulators (e.g., interferon) at enrollment or planned use during the study
* Receipt of any of the following: Prior use of emicizumab prophylaxis including investigational or commercial emicizumab; An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 drug-elimination half-lives of last drug administration; A non-hemophilia-related investigational drug within the last 30 days or 5 drug-elimination half-lives, whichever is shorter; An investigational drug concurrently
* Current active severe bleed, such as intracranial hemorrhage
* Planned surgery (excluding minor procedures, e.g., circumcision, CVAD placement) during the study
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Patients who are at high risk for thrombotic microangiopathy (TMA) (e.g., have a previous medical or family history of TMA, such as thrombotic thrombocytopenic purpura, atypical hemolytic uremic syndrome) in the investigator's judgment
* Previous or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis in patients for whom anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Any hereditary or acquired maternal condition that may predispose the patient to thrombotic events (e.g., inherited thrombophilias antiphospholipid syndrome)
* Other diseases (e.g., certain autoimmune diseases) that may increase risk of bleeding or thrombosis
* Known infection with HIV, hepatitis B virus, or hepatitis C virus
* Serious infection requiring antibiotics or antiviral treatments within 14 days prior to screening
* Concurrent disease, treatment, abnormality in clinical laboratory tests, vital signs measurements, or physical examination findings that could interfere with the conduct of the study or that would, in the opinion of the investigator or Sponsor, preclude the patient's safe participation in and completion of the study or interpretation of the study results
* Unwillingness of the parent or caregiver to allow receipt of blood or blood products, or any standard-of-care treatment for a life-threatening condition
* Any other medical, social, or other condition that may prevent adequate compliance with the study protocol in the opinion of the investigator

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2030-05-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Medizinische Universität Wien, Vienna, Austria
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Hospital das Clínicas Faculdades Médicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- Groupe Hospitalier Necker Enfants Malades, Paris, France
- Germany (2):
  - Universitätsklinikum Bonn, Bonn
  - Hämophilie-Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Sheba Medical Center - National Hemophilia Center, Tel Litwinsky, Israel
- Italy (4):
  - AORN Santobono Pausilipon, Napoli, Campania
  - AOU di Parma, Parma, Emilia-Romagna
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - AOU Careggi, Florence, Tuscany
- Charlotte Maxeke Johannesburg Hospital, Johannesburg, South Africa
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Turkey (Türkiye) (4):
  - Adana Acibadem Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Ege University, School of Medicine, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Pipe SW, Collins P, Dhalluin C, Kenet G, Schmitt C, Buri M, Jimenez-Yuste V, Peyvandi F, Young G, Oldenburg J, Mancuso ME, Kavakli K, Kiialainen A, Deb S, Niggli M, Chang T, Lehle M, Fijnvandraat K. Emicizumab prophylaxis in infants with hemophilia A (HAVEN 7): primary analysis of a phase 3b open-label trial. Blood. 2024 Apr 4;143(14):1355-1364. doi: 10.1182/blood.2023021832. PMID 38127586
- [Derived] Lopez-Jaime FJ, Benitez O, Diaz Jordan BL, Montano A, Coll J, Quintana Paris L, Gomez-Del Castillo Solano MDC. Expert opinion paper on the treatment of hemophilia a with emicizumab. Hematology. 2023 Dec;28(1):2166334. doi: 10.1080/16078454.2023.2166334. PMID 36636993
- [Derived] Hart DP. Commentary on "Development of a novel fully functional coagulation factor VIII with reduced immunogenicity utilizing an in silico prediction and deimmunization approach" - Will we ever be able to avoid inhibitor formation in hemophilia A? J Thromb Haemost. 2021 Sep;19(9):2125-2126. doi: 10.1111/jth.15404. No abstract available. PMID 34435432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 55 participants were enrolled in the study.
Groups:
- Emicizumab: Initially, all participants received loading doses of 3 milligrams per kilogram (mg/kg) emicizumab subcutaneously (SC) once every week (QW) for 4 weeks followed by the maintenance dosing regimen 3 mg/kg emicizumab SC once every 2 weeks (Q2W) for a total of 52 weeks. At the Week 53 clinic visit following consultation with the treating physician, parents/caregivers could have elected for their child to continue with the maintenance 3-mg/kg SC Q2W dosing regimen or to switch to the maintenance 1.5-mg/kg SC QW or 6-mg/kg SC once every 4 weeks (Q4W) dosing regimen for the subsequent 7-year long-term follow-up period.
Period: Overall Study
Arm/Group | Emicizumab
Started | 55
Received at Least One Dose of Study Drug (Safety Population) | 55
Completed 52 Weeks in the Study | 55
Started the Long-Term Follow-Up Period | 55
Completed | 0
Not Completed | 55
Not completed — Ongoing in the Study | 55

BASELINE CHARACTERISTICS:
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Months] | 5.0 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 48
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Annualized Bleeding Rate for Treated Bleeds
Description: The number of treated bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: From first dose of emicizumab to the clinical cutoff date or withdrawal date, whichever was earlier (median [range, min-max] efficacy period: 101.9 [52.6-119.7] weeks)
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated bleeds per year | 0.4 [0.30 to 0.63]

2. Primary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Bleeds
Description: The number of treated bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated bleed was defined as a bleed that was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated bleeds per year | 0.5 [0.00 to 4.59]

3. Primary Outcome: Median Calculated Annualized Bleeding Rate for Treated Bleeds
Description: as for outcome 2
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated bleeds per year | 0.0 [0.00 to 0.81]

4. Primary Outcome: Model-Based Annualized Bleeding Rate for All Bleeds
Description: The number of all bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
All bleeds per year | 2.0 [1.49 to 2.66]

5. Primary Outcome: Mean Calculated Annualized Bleeding Rate for All Bleeds
Description: The number of all bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule meant that two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: All bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
All bleeds per year | 2.0 [0.24 to 7.22]

6. Primary Outcome: Median Calculated Annualized Bleeding Rate for All Bleeds
Description: as for outcome 5
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: All bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
All bleeds per year | 1.0 [0.53 to 2.93]

7. Primary Outcome: Model-Based Annualized Bleeding Rate for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period was estimated as an annualized bleeding rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated spontaneous bleed was defined as a treated bleed (bleed directly followed by a hemophilia medication reported to be a "treatment for bleed") with no other known contributing factor such as trauma or procedure/surgery. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated spontaneous bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated spontaneous bleeds per year | NA [NA to NA] — No participants experienced treated spontaneous bleeds while receiving emicizumab prophylaxis up to the clinical cutoff date; thus, the ABR and 95% confidence interval could not be estimated using the model-based approach.

8. Primary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Spontaneous Bleeds
Description: The number of treated spontaneous bleeds over the efficacy period is presented here as a calculated annualized bleeding rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated spontaneous bleed was defined as a treated bleed (bleed directly followed by a hemophilia medication reported to be a "treatment for bleed") with no other known contributing factor such as trauma or procedure/surgery. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated spontaneous bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated spontaneous bleeds per year | 0.0 [NA to 3.69] — The lower limit of the 95% confidence interval could not be calculated because no participants experienced treated spontaneous bleeds up to the clinical cutoff date.

9. Primary Outcome: Median Calculated Annualized Bleeding Rate for Treated Spontaneous Bleeds
Description: as for outcome 8
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated spontaneous bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated spontaneous bleeds per year | 0.0 [0.00 to 0.00]

10. Primary Outcome: Model-Based Annualized Bleeding Rate for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period was estimated as an annualized bleed rate (ABR) using a negative binomial regression model, which accounts for different follow-up times. A treated joint bleed was defined as a bleed with type reported as "joint" based on at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline, and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Number (95% Confidence Interval); unit: Treated joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated joint bleeds per year | 0.0 [0.0 to 0.1]

11. Primary Outcome: Mean Calculated Annualized Bleeding Rate for Treated Joint Bleeds
Description: The number of treated joint bleeds over the efficacy period is presented here as a calculated annualized bleed rate (ABR) that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A treated joint bleed was defined as a bleed with type reported as "joint" based on at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline, and the bleed was directly followed by a hemophilia medication reported to be a "treatment for bleed". The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location were counted as one bleed if the second bleed occurred within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure were excluded.
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Mean (95% Confidence Interval); unit: Treated joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated joint bleeds per year | 0.0 [0.00 to 3.75]

12. Primary Outcome: Median Calculated Annualized Bleeding Rate for Treated Joint Bleeds
Description: as for outcome 11
Time Frame: as for outcome 1
Population: The Treated Population includes all participants who received at least one dose of emicizumab.
Measure: Median (Inter-Quartile Range); unit: Treated joint bleeds per year
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Treated joint bleeds per year | 0.0 [0.00 to 0.00]

13. Secondary Outcome: Hemophilia Joint Health Score (HJHS) Total Score at Specified Timepoints During the Long-Term Follow-Up Period
Time Frame: At Years 4, 5, 6, 7, and 8 of follow-up
Reporting Status: Not Posted, anticipated posting 2031-05

14. Secondary Outcome: Magnetic Resonance Imaging (MRI) Score of Specific Joints at Specified Timepoints During the Long-Term Follow-Up Period
Time Frame: At Years 5 and 8 of follow-up
Reporting Status: Not Posted, anticipated posting 2031-05

15. Secondary Outcome: Incidence and Severity of Adverse Events, With Severity Determined According to World Health Organization (WHO) Toxicity Grading Scale
Time Frame: From first dose of emicizumab until study completion (8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

16. Secondary Outcome: Incidence of Thromboembolic Events
Time Frame: From first dose of emicizumab until study completion (8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

17. Secondary Outcome: Incidence of Thrombotic Microangiopathy
Time Frame: From first dose of emicizumab until study completion (8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

18. Secondary Outcome: Incidence and Severity of of Injection Site Reactions, With Severity Determined According to WHO Toxicity Grading Scale
Time Frame: From first dose of emicizumab until study completion (8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

19. Secondary Outcome: Incidence of Severe Hypersensitivity, Anaphylaxis, and Anaphylactoid Events
Time Frame: From first dose of emicizumab until study completion (8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

20. Secondary Outcome: Incidence of Adverse Events Leading to Study Drug Discontinuation
Time Frame: From first dose of emicizumab until study completion (8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

21. Secondary Outcome: Number of Participants According to Hematology and Serum Chemistry Laboratory Test Result Shifts From Baseline WHO Grade to the Highest WHO Grade Post-Baseline
Description: Laboratory parameters for hematology and blood chemistry were measured at baseline and over time, and the values were compared with a standard reference range. Values outside the standard reference range were considered laboratory abnormalities and graded according to the World Health Organization (WHO) toxicity grading scale, ranging from lowest (Grade 1) to greatest (Grade 4) deviation from standard in the direction indicated for the abnormality (i.e., below (Low) or above (High) the reference range; 'Not Low' and 'Not High' indicate values within the reference range). Participants were categorized according to their laboratory test result shift from baseline WHO grade to highest WHO grade at any point post-baseline (up to Week 53) for each parameter. 'Missing' indicates that the test result was not available.
Time Frame: Baseline, Weeks 4, 13, 21, 29, 37, 45, and 53
Population: The Safety-Evaluable Population includes all participants who received at least one dose of emicizumab. The number analyzed (denominator) represents the total number of participants according to their baseline test result WHO toxicity grade for each parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
Participants
  Hemoglobin (Low), Not Low to Not Low: number analyzed (Participants) | 46
  Hemoglobin (Low), Not Low to Not Low | 36
  Hemoglobin (Low), Not Low to Grade 1: number analyzed (Participants) | 46
  Hemoglobin (Low), Not Low to Grade 1 | 5
  Hemoglobin (Low), Not Low to Grade 2: number analyzed (Participants) | 46
  Hemoglobin (Low), Not Low to Grade 2 | 5
  Hemoglobin (Low), Grade 1 to Not Low: number analyzed (Participants) | 8
  Hemoglobin (Low), Grade 1 to Not Low | 3
  Hemoglobin (Low), Grade 1 to Grade 1: number analyzed (Participants) | 8
  Hemoglobin (Low), Grade 1 to Grade 1 | 3
  Hemoglobin (Low), Grade 1 to Grade 3: number analyzed (Participants) | 8
  Hemoglobin (Low), Grade 1 to Grade 3 | 1
  Hemoglobin (Low), Grade 1 to Grade 4: number analyzed (Participants) | 8
  Hemoglobin (Low), Grade 1 to Grade 4 | 1
  Hemoglobin (Low), Grade 2 to Grade 2: number analyzed (Participants) | 1
  Hemoglobin (Low), Grade 2 to Grade 2 | 1
  Neutrophils, Total, Abs. (Low), Not Low to Not Low: number analyzed (Participants) | 29
  Neutrophils, Total, Abs. (Low), Not Low to Not Low | 8
  Neutrophils, Total, Abs. (Low), Not Low to Grade 1: number analyzed (Participants) | 29
  Neutrophils, Total, Abs. (Low), Not Low to Grade 1 | 14
  Neutrophils, Total, Abs. (Low), Not Low to Grade 2: number analyzed (Participants) | 29
  Neutrophils, Total, Abs. (Low), Not Low to Grade 2 | 2
  Neutrophils, Total, Abs. (Low), Not Low to Grade 3: number analyzed (Participants) | 29
  Neutrophils, Total, Abs. (Low), Not Low to Grade 3 | 3
  Neutrophils, Total, Abs. (Low), Not Low to Grade 4: number analyzed (Participants) | 29
  Neutrophils, Total, Abs. (Low), Not Low to Grade 4 | 2
  Neutrophils, Total, Abs. (Low), Grade 1 to Not Low: number analyzed (Participants) | 17
  Neutrophils, Total, Abs. (Low), Grade 1 to Not Low | 4
  Neutrophils, Total, Abs. (Low), Grade 1 to Grade 1: number analyzed (Participants) | 17
  Neutrophils, Total, Abs. (Low), Grade 1 to Grade 1 | 7
  Neutrophils, Total, Abs. (Low), Grade 1 to Grade 2: number analyzed (Participants) | 17
  Neutrophils, Total, Abs. (Low), Grade 1 to Grade 2 | 5
  Neutrophils, Total, Abs. (Low), Grade 1 to Grade 3: number analyzed (Participants) | 17
  Neutrophils, Total, Abs. (Low), Grade 1 to Grade 3 | 1
  Neutrophils, Total, Abs. (Low), Grade 2 to Not Low: number analyzed (Participants) | 5
  Neutrophils, Total, Abs. (Low), Grade 2 to Not Low | 1
  Neutrophils, Total, Abs. (Low), Grade 2 to Grade 1: number analyzed (Participants) | 5
  Neutrophils, Total, Abs. (Low), Grade 2 to Grade 1 | 2
  Neutrophils, Total, Abs. (Low), Grade 2 to Grade 2: number analyzed (Participants) | 5
  Neutrophils, Total, Abs. (Low), Grade 2 to Grade 2 | 1
  Neutrophils, Total, Abs. (Low), Grade 2 to Grade 3: number analyzed (Participants) | 5
  Neutrophils, Total, Abs. (Low), Grade 2 to Grade 3 | 1
  Neutrophils, Total, Abs. (Low), Missing to Not Low: number analyzed (Participants) | 3
  Neutrophils, Total, Abs. (Low), Missing to Not Low | 1
  Neutrophils, Total, Abs. (Low), Missing to Grade 1: number analyzed (Participants) | 3
  Neutrophils, Total, Abs. (Low), Missing to Grade 1 | 1
  Neutrophils, Total, Abs. (Low), Missing to Grade 2: number analyzed (Participants) | 3
  Neutrophils, Total, Abs. (Low), Missing to Grade 2 | 1
  Platelets (Low), Not Low to Not Low | 54
  Platelets (Low), Not Low to Grade 2 | 1
  Alkaline Phosphatase (High), Not High to Not High: number analyzed (Participants) | 44
  Alkaline Phosphatase (High), Not High to Not High | 32
  Alkaline Phosphatase (High), Not High to Grade 1: number analyzed (Participants) | 44
  Alkaline Phosphatase (High), Not High to Grade 1 | 6
  Alkaline Phosphatase (High), Not High to Grade 2: number analyzed (Participants) | 44
  Alkaline Phosphatase (High), Not High to Grade 2 | 2
  Alkaline Phosphatase (High), Not High to Grade 3: number analyzed (Participants) | 44
  Alkaline Phosphatase (High), Not High to Grade 3 | 1
  Alkaline Phosphatase (High), Not High to Grade 4: number analyzed (Participants) | 44
  Alkaline Phosphatase (High), Not High to Grade 4 | 3
  Alkaline Phosphatase (High), Grade 1 to Not High: number analyzed (Participants) | 6
  Alkaline Phosphatase (High), Grade 1 to Not High | 2
  Alkaline Phosphatase (High), Grade 1 to Grade 1: number analyzed (Participants) | 6
  Alkaline Phosphatase (High), Grade 1 to Grade 1 | 3
  Alkaline Phosphatase (High), Grade 1 to Grade 3: number analyzed (Participants) | 6
  Alkaline Phosphatase (High), Grade 1 to Grade 3 | 1
  Alkaline Phosphatase (High), Grade 2 to Not High: number analyzed (Participants) | 3
  Alkaline Phosphatase (High), Grade 2 to Not High | 1
  Alkaline Phosphatase (High), Grade 2 to Grade 1: number analyzed (Participants) | 3
  Alkaline Phosphatase (High), Grade 2 to Grade 1 | 1
  Alkaline Phosphatase (High), Grade 2 to Grade 2: number analyzed (Participants) | 3
  Alkaline Phosphatase (High), Grade 2 to Grade 2 | 1
  Alkaline Phosphatase (High), Missing to Not High: number analyzed (Participants) | 2
  Alkaline Phosphatase (High), Missing to Not High | 1
  Alkaline Phosphatase (High), Missing to Grade 1: number analyzed (Participants) | 2
  Alkaline Phosphatase (High), Missing to Grade 1 | 1
  SGPT/ALT (High), Not High to Not High: number analyzed (Participants) | 51
  SGPT/ALT (High), Not High to Not High | 43
  SGPT/ALT (High), Not High to Grade 1: number analyzed (Participants) | 51
  SGPT/ALT (High), Not High to Grade 1 | 6
  SGPT/ALT (High), Not High to Grade 3: number analyzed (Participants) | 51
  SGPT/ALT (High), Not High to Grade 3 | 1
  SGPT/ALT (High), Not High to Grade 4: number analyzed (Participants) | 51
  SGPT/ALT (High), Not High to Grade 4 | 1
  SGPT/ALT (High), Grade 1 to Grade 1: number analyzed (Participants) | 3
  SGPT/ALT (High), Grade 1 to Grade 1 | 2
  SGPT/ALT (High), Grade 1 to Grade 4: number analyzed (Participants) | 3
  SGPT/ALT (High), Grade 1 to Grade 4 | 1
  SGPT/ALT (High), Missing to Not High: number analyzed (Participants) | 1
  SGPT/ALT (High), Missing to Not High | 1
  SGOT/AST (High), Not High to Not High: number analyzed (Participants) | 44
  SGOT/AST (High), Not High to Not High | 31
  SGOT/AST (High), Not High to Grade 1: number analyzed (Participants) | 44
  SGOT/AST (High), Not High to Grade 1 | 11
  SGOT/AST (High), Not High to Grade 3: number analyzed (Participants) | 44
  SGOT/AST (High), Not High to Grade 3 | 2
  SGOT/AST (High), Grade 1 to Not High: number analyzed (Participants) | 11
  SGOT/AST (High), Grade 1 to Not High | 2
  SGOT/AST (High), Grade 1 to Grade 1: number analyzed (Participants) | 11
  SGOT/AST (High), Grade 1 to Grade 1 | 8
  SGOT/AST (High), Grade 1 to Grade 3: number analyzed (Participants) | 11
  SGOT/AST (High), Grade 1 to Grade 3 | 1
  Blood Urea Nitrogen (High), Not High to Not High: number analyzed (Participants) | 47
  Blood Urea Nitrogen (High), Not High to Not High | 42
  Blood Urea Nitrogen (High), Not High to Grade 1: number analyzed (Participants) | 47
  Blood Urea Nitrogen (High), Not High to Grade 1 | 5
  Blood Urea Nitrogen (High), Grade 1 to Grade 1: number analyzed (Participants) | 2
  Blood Urea Nitrogen (High), Grade 1 to Grade 1 | 2
  Blood Urea Nitrogen (High), Missing to Not High: number analyzed (Participants) | 4
  Blood Urea Nitrogen (High), Missing to Not High | 4
  Calcium (High), Not High to Not High: number analyzed (Participants) | 31
  Calcium (High), Not High to Not High | 13
  Calcium (High), Not High to Grade 1: number analyzed (Participants) | 31
  Calcium (High), Not High to Grade 1 | 18
  Calcium (High), Grade 1 to Not High: number analyzed (Participants) | 20
  Calcium (High), Grade 1 to Not High | 2
  Calcium (High), Grade 1 to Grade 1: number analyzed (Participants) | 20
  Calcium (High), Grade 1 to Grade 1 | 17
  Calcium (High), Grade 1 to Grade 2: number analyzed (Participants) | 20
  Calcium (High), Grade 1 to Grade 2 | 1
  Calcium (High), Grade 2 to Grade 1: number analyzed (Participants) | 1
  Calcium (High), Grade 2 to Grade 1 | 1
  Calcium (High), Missing to Not High: number analyzed (Participants) | 3
  Calcium (High), Missing to Not High | 3
  Calcium, Corrected for Albumin (High), Not High to Not High: number analyzed (Participants) | 38
  Calcium, Corrected for Albumin (High), Not High to Not High | 32
  Calcium, Corrected for Albumin (High), Not High to Grade 1: number analyzed (Participants) | 38
  Calcium, Corrected for Albumin (High), Not High to Grade 1 | 6
  Calcium, Corrected for Albumin (High), Grade 1 to Not High: number analyzed (Participants) | 11
  Calcium, Corrected for Albumin (High), Grade 1 to Not High | 6
  Calcium, Corrected for Albumin (High), Grade 1 to Grade 1: number analyzed (Participants) | 11
  Calcium, Corrected for Albumin (High), Grade 1 to Grade 1 | 5
  Calcium, Corrected for Albumin (High), Missing to Not High: number analyzed (Participants) | 6
  Calcium, Corrected for Albumin (High), Missing to Not High | 5
  Calcium, Corrected for Albumin (High), Missing to Grade 1: number analyzed (Participants) | 6
  Calcium, Corrected for Albumin (High), Missing to Grade 1 | 1
  Creatinine (High), Not High to Not High | 53
  Creatinine (High), Not High to Grade 1 | 2
  Glucose (High), Not High to Not High: number analyzed (Participants) | 52
  Glucose (High), Not High to Not High | 51
  Glucose (High), Not High to Grade 1: number analyzed (Participants) | 52
  Glucose (High), Not High to Grade 1 | 1
  Glucose (High), Missing to Not High: number analyzed (Participants) | 3
  Glucose (High), Missing to Not High | 3
  Potassium (High), Not High to Not High: number analyzed (Participants) | 47
  Potassium (High), Not High to Not High | 40
  Potassium (High), Not High to Grade 1: number analyzed (Participants) | 47
  Potassium (High), Not High to Grade 1 | 7
  Potassium (High), Grade 1 to Not High: number analyzed (Participants) | 5
  Potassium (High), Grade 1 to Not High | 4
  Potassium (High), Grade 1 to Grade 3: number analyzed (Participants) | 5
  Potassium (High), Grade 1 to Grade 3 | 1
  Potassium (High), Missing to Not High: number analyzed (Participants) | 3
  Potassium (High), Missing to Not High | 1
  Potassium (High), Missing to Grade 1: number analyzed (Participants) | 3
  Potassium (High), Missing to Grade 1 | 1
  Potassium (High), Missing to Grade 3: number analyzed (Participants) | 3
  Potassium (High), Missing to Grade 3 | 1
  Sodium (High), Not High to Not High: number analyzed (Participants) | 52
  Sodium (High), Not High to Not High | 52
  Sodium (High), Grade 1 to Not High: number analyzed (Participants) | 1
  Sodium (High), Grade 1 to Not High | 1
  Sodium (High), Missing to Not High: number analyzed (Participants) | 2
  Sodium (High), Missing to Not High | 2
  Bilirubin (High), Not High to Not High: number analyzed (Participants) | 44
  Bilirubin (High), Not High to Not High | 43
  Bilirubin (High), Not High to Grade 1: number analyzed (Participants) | 44
  Bilirubin (High), Not High to Grade 1 | 1
  Bilirubin (High), Grade 1 to Not High: number analyzed (Participants) | 1
  Bilirubin (High), Grade 1 to Not High | 1
  Bilirubin (High), Grade 2 to Not High: number analyzed (Participants) | 3
  Bilirubin (High), Grade 2 to Not High | 3
  Bilirubin (High), Grade 3 to Not High: number analyzed (Participants) | 3
  Bilirubin (High), Grade 3 to Not High | 2
  Bilirubin (High), Grade 3 to Grade 1: number analyzed (Participants) | 3
  Bilirubin (High), Grade 3 to Grade 1 | 1
  Bilirubin (High), Grade 4 to Not High: number analyzed (Participants) | 4
  Bilirubin (High), Grade 4 to Not High | 1
  Bilirubin (High), Grade 4 to Grade 2: number analyzed (Participants) | 4
  Bilirubin (High), Grade 4 to Grade 2 | 1
  Bilirubin (High), Grade 4 to Grade 3: number analyzed (Participants) | 4
  Bilirubin (High), Grade 4 to Grade 3 | 2
  Calcium (Low), Not Low to Not Low: number analyzed (Participants) | 52
  Calcium (Low), Not Low to Not Low | 50
  Calcium (Low), Not Low to Grade 4: number analyzed (Participants) | 52
  Calcium (Low), Not Low to Grade 4 | 2
  Calcium (Low), Missing to Not Low: number analyzed (Participants) | 3
  Calcium (Low), Missing to Not Low | 3
  Calcium, Corrected for Albumin (Low), Not Low to Not Low: number analyzed (Participants) | 49
  Calcium, Corrected for Albumin (Low), Not Low to Not Low | 47
  Calcium, Corrected for Albumin (Low), Not Low to Grade 4: number analyzed (Participants) | 49
  Calcium, Corrected for Albumin (Low), Not Low to Grade 4 | 2
  Calcium, Corrected for Albumin (Low), Missing to Not Low: number analyzed (Participants) | 6
  Calcium, Corrected for Albumin (Low), Missing to Not Low | 6
  Glucose (Low), Not Low to Not Low: number analyzed (Participants) | 51
  Glucose (Low), Not Low to Not Low | 44
  Glucose (Low), Not Low to Grade 1: number analyzed (Participants) | 51
  Glucose (Low), Not Low to Grade 1 | 6
  Glucose (Low), Not Low to Grade 2: number analyzed (Participants) | 51
  Glucose (Low), Not Low to Grade 2 | 1
  Glucose (Low), Grade 1 to Not Low: number analyzed (Participants) | 1
  Glucose (Low), Grade 1 to Not Low | 1
  Glucose (Low), Missing to Not Low: number analyzed (Participants) | 3
  Glucose (Low), Missing to Not Low | 3
  Magnesium (Low), Not Low to Not Low: number analyzed (Participants) | 50
  Magnesium (Low), Not Low to Not Low | 50
  Magnesium (Low), Grade 1 to Not Low: number analyzed (Participants) | 2
  Magnesium (Low), Grade 1 to Not Low | 2
  Magnesium (Low), Missing to Not Low: number analyzed (Participants) | 3
  Magnesium (Low), Missing to Not Low | 3
  Phosphorus (Low), Not Low to Not Low: number analyzed (Participants) | 52
  Phosphorus (Low), Not Low to Not Low | 52
  Phosphorus (Low), Missing to Not Low: number analyzed (Participants) | 3
  Phosphorus (Low), Missing to Not Low | 3
  Postassium (Low), Not Low to Not Low: number analyzed (Participants) | 52
  Postassium (Low), Not Low to Not Low | 52
  Postassium (Low), Missing to Not Low: number analyzed (Participants) | 3
  Postassium (Low), Missing to Not Low | 3
  Sodium (Low), Not Low to Not Low: number analyzed (Participants) | 48
  Sodium (Low), Not Low to Not Low | 35
  Sodium (Low), Not Low to Grade 1: number analyzed (Participants) | 48
  Sodium (Low), Not Low to Grade 1 | 13
  Sodium (Low), Grade 1 to Not Low: number analyzed (Participants) | 5
  Sodium (Low), Grade 1 to Not Low | 1
  Sodium (Low), Grade 1 to Grade 1: number analyzed (Participants) | 5
  Sodium (Low), Grade 1 to Grade 1 | 4
  Sodium (Low), Missing to Not Low: number analyzed (Participants) | 2
  Sodium (Low), Missing to Not Low | 1
  Sodium (Low), Missing to Grade 1: number analyzed (Participants) | 2
  Sodium (Low), Missing to Grade 1 | 1

22. Secondary Outcome: Change From Baseline in Pulse Rate Over Time
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53, and annually during the 7-year follow-up period until study completion (up to 8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

23. Secondary Outcome: Change From Baseline in Respiratory Rate Over Time
Time Frame: as for outcome 22
Reporting Status: Not Posted, anticipated posting 2031-05

24. Secondary Outcome: Change From Baseline in Body Temperature Over Time
Time Frame: as for outcome 22
Reporting Status: Not Posted, anticipated posting 2031-05

25. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Time Frame: as for outcome 22
Reporting Status: Not Posted, anticipated posting 2031-05

26. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Time Frame: as for outcome 22
Reporting Status: Not Posted, anticipated posting 2031-05

27. Secondary Outcome: Plasma Trough Concentrations (Ctrough) of Emicizumab
Time Frame: Predose at Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: The Pharmacokinetic (PK)-Evaluable Population: includes all participants who had received at least one dose of emicizumab and had at least one post-baseline emicizumab plasma concentration result. The number analyzed indicates the number of participants who provided a PK sample at a given timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Emicizumab
Number analyzed (Participants) | 55
micrograms per millilitre (μg/mL)
  Week 1: number analyzed (Participants) | 50
  Week 1 | NA (NA) — The mean and standard deviation could not be calculated because all samples were below the limit of quantitation. The samples were taken prior to administration of the first dose.
  Week 3: number analyzed (Participants) | 51
  Week 3 | 36.8 (9.8)
  Week 5: number analyzed (Participants) | 52
  Week 5 | 62.0 (13.4)
  Week 7: number analyzed (Participants) | 51
  Week 7 | 62.3 (13.5)
  Week 9: number analyzed (Participants) | 51
  Week 9 | 64.2 (14.4)
  Week 13: number analyzed (Participants) | 52
  Week 13 | 66.0 (12.0)
  Week 17: number analyzed (Participants) | 51
  Week 17 | 65.8 (13.1)
  Week 21: number analyzed (Participants) | 49
  Week 21 | 65.8 (13.9)
  Week 25: number analyzed (Participants) | 52
  Week 25 | 65.6 (15.1)
  Week 29: number analyzed (Participants) | 53
  Week 29 | 63.2 (14.6)
  Week 33: number analyzed (Participants) | 50
  Week 33 | 64.0 (21.5)
  Week 37: number analyzed (Participants) | 50
  Week 37 | 63.1 (15.8)
  Week 41: number analyzed (Participants) | 48
  Week 41 | 62.0 (17.6)
  Week 45: number analyzed (Participants) | 52
  Week 45 | 59.9 (16.6)
  Week 49: number analyzed (Participants) | 52
  Week 49 | 57.1 (14.7)
  Week 53: number analyzed (Participants) | 52
  Week 53 | 56.8 (15.3)

28. Secondary Outcome: Incidence of Anti-Emicizumab Antibodies
Time Frame: Weeks 1, 5, 17, 29, 41, and 53, and thereafter as clinically indicated until study completion (up to 8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

29. Secondary Outcome: Incidence of De Novo Development of Factor VIII Inhibitors
Description: As per the protocol, after any 3 exposure days to FVIII or a block of FVIII exposure days (e.g., a block is defined as a minimum of two consecutive doses of FVIII) administered for treatment of a bleed, a surgical procedure, or other (e.g., preventative doses before activity), one plasma sample for anti-FVIII antibodies (for centralized analysis) had to be collected 14 days after the final dose of FVIII administered.
Time Frame: As clinically indicated from baseline until study completion (up to 8 years)
Reporting Status: Not Posted, anticipated posting 2031-05

ADVERSE EVENTS:
Time Frame: From first dose of emicizumab until the primary completion date cutoff (median [range, min-max] observation period: 101.9 [52.6-119.7] weeks)
Description: Adverse events (AEs) are reported in the Safety-Evaluable/Treated Population, comprising all participants who received at least one dose of emicizumab. AEs are still being collected until the end of the study and the results will be updated within 1 year of the date of final data collection.
Arm/Group | Emicizumab
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 16/55
Other Adverse Events (participants affected / at risk) | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emicizumab (N=55)
Bronchiolitis (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 3 (4)
Eyelid contusion (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2)
Tongue haemorrhage (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emicizumab (N=55)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (14)
Teething (Gastrointestinal disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 8 (11)
Constipation (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 26 (51)
Injection site reaction (General disorders) | 11 (32)
Hyperpyrexia (General disorders) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 22 (57)
Nasopharyngitis (Infections and infestations) | 18 (39)
COVID-19 (Infections and infestations) | 16 (16)
Bronchitis (Infections and infestations) | 8 (8)
Ear infection (Infections and infestations) | 7 (15)
Gastroenteritis (Infections and infestations) | 8 (12)
Conjunctivitis (Infections and infestations) | 7 (10)
Viral upper respiratory tract infection (Infections and infestations) | 7 (16)
Viral infection (Infections and infestations) | 5 (10)
Hand-foot-and-mouth disease (Infections and infestations) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 4 (5)
Otitis media (Infections and infestations) | 4 (5)
Gastrointestinal infection (Infections and infestations) | 3 (3)
Varicella (Infections and infestations) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 16 (32)
Head injury (Injury, poisoning and procedural complications) | 10 (18)
Rash (Skin and subcutaneous tissue disorders) | 10 (11)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (20)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 3 (4)
Iron deficiency (Metabolism and nutrition disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT04431726/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT04431726/SAP_001.pdf